CLINICAL TRIAL: NCT07227974
Title: Empower EI: Comparing Early Intervention Approaches to Improve Communication in Toddlers With Developmental Delays
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPS-2024C1-38924
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Developmental Delays
Keywords: Developmental Disabilities; Language Delay; Caregiver Coaching; Caregiver Responsiveness; Early Intervention; Pragmatic Clinical Trial; Communication; Speech-Language Pathology; Patient-Centered Outcomes Research
MeSH Terms: conditions — Developmental Disabilities; Language Development Disorders; Communication

STUDY DESIGN:
Intervention Model Description: This is a three-arm randomized controlled trial designed to compare the effectiveness of different approaches to Early Intervention (EI) service delivery for toddlers with speech and communication delays. Participants will be randomly assigned to one of three intervention models
  Each approach will be delivered over a 28-week period, with evaluations occurring at baseline, 14 and 28 weeks. The study will assess child outcomes (e.g., social communication) and caregiver outcomes (e.g., use of responsive strategies and capacity to support their child's needs).
  Participants will be randomized within their Early Intervention speech therapist, with stratification by race.
  This randomized design enables direct comparisons across intervention models to determine which approaches are most effective for different families and to identify factors that influence their effectiveness.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapist-Delivered Early Intervention Approach (Active Comparator): For 28 weeks, this arm will receive the therapist-delivered early intervention approach.
  Interventions: Behavioral: Therapist-Delivered Early Intervention Approach
- Caregiver Coaching Early Intervention Approach (Experimental): For 28 weeks, this arm will receive the caregiver coaching early intervention approach.
  Interventions: Behavioral: Caregiver Coaching Early Intervention Approach
- Combined Early Intervention Approach + Parents Taking Action (Experimental): For the first 14 weeks, this arm will receive the therapist-delivered early intervention as well as Parents Taking Action. For the following 14 weeks, this arm will receive the caregiver coaching early intervention approach.
  Interventions: Behavioral: Therapist-Delivered Early Intervention Approach; Behavioral: Caregiver Coaching Early Intervention Approach; Behavioral: Parents Taking Action

INTERVENTIONS:
Behavioral: Therapist-Delivered Early Intervention Approach — The therapist-delivered early intervention approach will occur during the child's weekly, hour-long early intervention (EI) sessions. During the sessions, the child's EI speech-language pathologist (SLP) will use responsive strategies directly with the child. Responsive strategies focus on noticing the child's communication and responding with language related to their focus of attention. The SLP will not coach the caregiver during the sessions.
  Arms: Combined Early Intervention Approach + Parents Taking Action; Therapist-Delivered Early Intervention Approach
Behavioral: Caregiver Coaching Early Intervention Approach — The caregiver-coaching early intervention approach will occur during the child's weekly, hour-long early intervention (EI) sessions. During the sessions, the child's EI speech-language pathologist (SLP) will coach the caregiver to use responsive strategies with their child. Responsive strategies focus on noticing the child's communication and responding with language related to their focus of attention.
  Arms: Caregiver Coaching Early Intervention Approach; Combined Early Intervention Approach + Parents Taking Action
Behavioral: Parents Taking Action — Parents Taking Action (PTA) will be delivered during weekly, one-hour virtual sessions with the caregiver, separate from the child's early intervention (EI) sessions. PTA is a psychoeducation program implemented by a peer mentor (i.e., a culturally-matched caregiver of a child with a developmental disability). During the sessions, the peer mentor will provide information and guidance on a range of topics (e.g., child development, early intervention systems, special education rights/resources, and advocacy) following a structured curriculum.
  Arms: Combined Early Intervention Approach + Parents Taking Action

SUMMARY:
This study is testing three ways to deliver Early Intervention (EI) services for toddlers with developmental disabilities (DD).

Children enrolled in EI speech therapy will receive one of three approaches:

1. Therapist Delivered EI: For 28 weeks, the child's speech therapist will work directly with the child to support their communication.
2. Caregiver Coaching EI: For 28 weeks, the child's speech therapist will coach the caregiver on how to support their child's communication.
3. Combined EI Approach + Parent-Led Education Program: For 14 weeks, the caregiver will take part in a parent-led education program while the speech therapist works directly with the child to support their communication. During the next 14 weeks, the speech therapist will coach the caregiver on how to support their child's communication.

The goal of this study is to identify which approaches are most effective so that all families can benefit fully from EI services.

DETAILED DESCRIPTION:
High-quality Early Intervention (EI) during the first three years of life, a period of heightened neuroplasticity, is critical to improving outcomes for children with developmental disabilities (DD). There are two EI approaches that may be effective for supporting child communication and improving family outcomes: 1) caregiver coaching, in which the EI therapist teaches the caregiver strategies to help their child's communication, and 2) caregiver psychoeducation, in which a peer mentor teaches the caregiver about skills and resources that are helpful in supporting their child and family.

The aim of the current clinical trial is to determine which EI approaches are most effective, for which families, and why they are effective. This clinical trial also aims to investigate how therapists are delivering the interventions and to characterize the acceptability and feasibility of these interventions for use in real-world settings.

A total of 1,269 toddlers (approximately equal numbers of Black, Latine, and white children) will be enrolled across community-based EI sites. Families will be directly recruited from participating EI therapists' existing caseloads. Caregiver-child dyads will be randomly assigned to one of three groups:

1. Therapist Delivered EI: For 28 weeks, the child's speech therapist will work directly with the child to support their communication.
2. Caregiver Coaching EI: For 28 weeks, the child's speech therapist will coach the caregiver on how to support their child's communication.
3. Combined EI Approach + Parents Taking Action: For 14 weeks, the caregiver will take part in a parent-led education program (Parents Taking Action) while the speech therapist works directly with the child to support their communication. During the next 14 weeks, the speech therapist will coach the caregiver on how to support their child's communication.

Outcomes will assess both caregiver and child domains, including caregiver use of responsive strategies, caregiver capacity to support the child's needs, and child social communication. The study will also examine moderators (e.g., race) and mediators (e.g., caregiver use of responsive strategies) to identify for whom and why each approach is most effective.

A process evaluation will assess implementation fidelity (quality, dosage, adaptations) and explore how fidelity influences effectiveness outcomes. Feasibility, acceptability, and appropriateness of each approach will be evaluated through surveys and interviews with caregivers and EI therapists.

This study is among the first large-scale comparative effectiveness trials of early intervention approaches conducted in real-world EI settings. Findings will inform EI practices and guide caregivers, therapists, and policymakers in selecting interventions that best meet the needs and preferences of diverse families.

ELIGIBILITY:
Child Inclusion Criteria:

* Age at enrollment: Older than 12 months and younger than 28 months
* Enrolled in the Illinois Early Intervention system and newly eligible for speech-language therapy (i.e., no prior EI speech-language therapy experience).
* Plans to receive one hour of speech-language therapy per week in the home or in a private space outside of the home

Child Exclusion Criteria

- Exposed to a language other than English or Spanish more than 10% of the time

Caregiver Inclusion Criteria:

* The child's parent, legal guardian, or other family member
* Self-identifies as Black, Latine (Hispanic), or white
* Available to participate in weekly EI sessions and study assessments.

Caregiver Exclusion Criteria

* Younger than 18 years old at enrollment
* Uses a language other than English or Spanish during their interactions with the child more than 10% of the time

Ages: 12 Months to 28 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1269 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Responsive Strategy Use (RSU) Rating Scale | Week 14, Week 28
  The Responsive Strategy Use (RSU) Rating Scale will be used to measure caregivers' use of responsive strategies during a naturalistic, caregiver-child interaction. Items on the RSU Rating Scale are rated on a 5-point Likert Scale (1 = Novice, 5 = Expert) and averaged to yield the RSU Total Score (Min = 1, Max = 5), with higher scores reflecting a stronger proficiency of responsive strategy use.
Family Outcomes Survey - Revised | Week 14, Week 28
  The Family Outcomes Survey-Revised is a 24-item informant-report questionnaire that assesses caregivers' understanding, confidence, and ability to support their child's needs. The Family Outcomes Total Score (Min = 24, Max = 120) reflects the caregiver's capacity to support their child's needs, with higher scores indicating greater capacity.
Communication and Symbolic Behavior Scales - Developmental Profile (CSBS-DP) | Week 28
  The Communication and Symbolic Behavior Scales - Developmental Profile (CSBS-DP) is a structured, norm-referenced, observational measure of child communication. The assessment is scored for 20 items across 7 domains (i.e., Emotion and Eye Gaze, Communication, Gestures, Sounds, Words, Understanding, Object Use). The weighted raw scores for each of the 7 domains are grouped into 3 clusters (social, speech, and symbolic) and combined into a total raw score (min = 0; max = 113). Higher scores indicate better skills.

SECONDARY OUTCOMES:
Session Attendance | Week 1 to Week 28
  Session attendance will be documented in weekly session logs completed by interventionists and summarized as the percentage of planned intervention sessions attended by each family (Min = 0%, Max = 100%).
Intervention Fidelity Checklist | Week 1 to Week 28
  The Intervention Fidelity Checklist is a rating scale assessing adherence to the intervention protocol. Items on the checklist correspond to the core elements of the respective intervention protocol and are scored based on specific behavioral criteria. The Intervention Fidelity Checklist will be scored on a randomly selected 20% of intervention sessions per participant. Scores will be averaged across sessions to yield an average intervention quality score (Min = 0, Max = 100), with higher scores indicating higher intervention quality.
Framework for Reporting Adaptations and Modifications (FRAME) | Week 1 to Week 28
  The Framework for Reporting Adaptations and Modifications (FRAME) will be used to document intervention adaptations. After each intervention session, interventionists will record intervention adaptations in a session log, including what was changed, for whom, the type of modification, and the reason. These data will yield the total number of adaptations (Min = 0, Max = NA).

OTHER OUTCOMES:
Early Intervention Program Satisfaction Scale | Week 14, Week 28
  An adapted version of the Early Intervention Program Satisfaction Scale, a caregiver-report questionnaire, will be used to assess caregiver satisfaction. This survey includes 6 items rated on a 5-point Likert (1 = Very Dissatisfied, 5 = Very Satisfied). The Total Score (Min = 6, Max = 30) reflects caregivers' overall satisfaction with the intervention, with higher scores representing greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Roberts, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in any publication arising from this trial will be made publicly available via the Dryad repository. The shared dataset will include all variables necessary to reproduce the published findings, including treatment assignment, participant demographics, baseline characteristics, and outcome measures. All data will be de-identified in accordance with HIPAA standards and institutional policies to protect participant confidentiality.
  Data will be uploaded to Dryad after publication of the primary results, and will be freely accessible to qualified researchers without restriction. A corresponding DOI will be provided in publications to facilitate data access and citation.
Supporting Information: Analytic Code
Time Frame: Data will be uploaded to the Dryad data repository on November 1st, 2030 and remain there indefinitely.
Access Criteria: De-identified individual participant data (IPD) and supporting documentation (e.g., data dictionaries, survey instruments, codebooks) will be publicly available to any researcher or member of the public. All data will be uploaded to the Dryad Digital Repository, where users can freely access and download the datasets. No special request or application will be required to access the IPD. The data will be shared in a de-identified format to protect participant privacy, and users will be able to access the IPD along with associated documentation necessary to understand and use the data for secondary analyses or replication studies.